CLINICAL TRIAL: NCT02429570
Title: Pilot Study of Meclofenamate in Subjects With Recurrent or Progressive Brain Metastasis From Solid Tumor Primary
Brief Title: Meclofenamate in Subjects With Recurrent or Progressive Brain Metastasis From Solid Tumor Primary
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-068
Record Dates: First submitted 2015-04-22; First posted 2015-04-29 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Brain Metastases; Progressive Brain Metastases
Keywords: meclofenamate; 15-068
MeSH Terms: conditions — Brain Neoplasms | interventions — Meclofenamic Acid

ARMS (1):
- Meclofenamate (Experimental): All enrolled patients will receive the study drug, meclofenamate at 100 mg PO BID.
  Interventions: Drug: Meclofenamate

INTERVENTIONS:
Drug: Meclofenamate

SUMMARY:
Cancer that has spread to the brain, or brain metastasis, is difficult to treat. Meclofenamate is a drug which has been shown to reduce brain metastasis growth in the laboratory. This medicine has been used in the past to treat pain. But, in this study, it will be used to prevent new brain metastasis. This is the first time that meclofenamate will be used in patients with brain metastasis.

This is a pilot study which means that the purpose of this study is to determine if a larger clinical trial of meclofenamate is possible in patients with brain metastasis. This study also aims to find out what effects, good and/or bad meclofenamate has on the patient and the cancer that has spread to the brain. The investigators also want to learn more about potential effects that this drug may have in the digestive system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* KPS ≥ 60
* At least one recurrent or progressive brain metastasis (es) from any solid primary tumor that is visible on MRI as assessed by the patient's treating physician.
* Recurrence may occur after any treatment: recurrence after whole-brain radiation, stereotactic radiosurgery, surgical resection, systemic chemotherapy are all acceptable.
* There is no limit on the number of brain metastases.
* Surgical resection or SRS to other recurrent lesions in the same patient are acceptable, provided one recurrent lesion remains untreated.
* Systemic disease must be well-controlled or NED in the opinion of the patient's primary oncologist.

Exclusion Criteria:

* Inability to get brain MRI +/- contrast
* Progressive systemic disease
* Known leptomeningeal metastases
* Primary Brain tumor
* Active Intracranial Hemorrhage
* Surgery less than two weeks before enrollment
* GI hemorrhage (active or in recent 6 months)
* Concurrent anti-platelet therapy
* Concurrent anti-coagulation therapy
* Active bleeding diathesis
* Platelet count ≤ 70,000/mm3
* International normalized ratio (INR) > 1.6 and a Partial Thromboplastin Time (PTT) > 40 seconds
* Serum Creatinine >2 mg/dL OR CrCL <30ml/min
* AST or ALT > 200 U/L
* Hemoglobin <8 g/dL
* Allergy to meclofenamate or other NSAID
* Inability to tolerate PO dosing
* Steroid dose increased in the most recent two weeks.
* Pregnancy
* Cardiac Arrhythmia requiring medical management and/or pacemaker.
* Known congestive heart failure requiring medical management

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasible (if at least 50% of patients enrolled are evaluable in brain by MRI at the 2-month timepoint) | 2 month
  The trial will be deemed "feasible" if at least 50% of patients enrolled are evaluable in brain by MRI at the 2-month timepoint.

SECONDARY OUTCOMES:
Adverse events | 1 year
  Adverse events (from all categories) will be collected, graded according to version 4.0 of the NCI Common Terminology Criteria for Adverse Events.
Progression free survival | 1 year
  progression-free survival is defined as time from start of treatment to progressive disease by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Boire, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cance Center
Locations (7):
- United States (7):
  - Baptist Health South Florida, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- [Derived] Laghetti P, Saltarella I, Dell'Atti S, Desaphy JF, Altamura C. Pleiotropic Effects of the NSAID Fenamates on Chloride Channels: Opportunity for Ion Channelopathies? Pharmacol Res Perspect. 2025 Aug;13(4):e70144. doi: 10.1002/prp2.70144. PMID 40568930
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/